CLINICAL TRIAL: NCT03903965
Title: Comparison of Retinal Perfusion Between Diabetic and Non-diabetic Patients With OCT Angiography After Cataract Surgery.
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hong Qi, Principal Investigator, Peking University Third Hospital
Other Study IDs: 2019032501
Record Dates: First submitted 2019-03-26; First posted 2019-04-04 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus Type 2; Age Related Cataracts
Keywords: diabetes; OCT Angiography; cataract surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — aqueous humor from the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic patients after cataract surgery: diabetic patients after cataract surgery
- non-diabetic patients after cataract surgery: non-diabetic patients after cataract surgery

SUMMARY:
This study aims to compare the retinal perfusion between diabetic and non-diabetic patients with Optical Coherence Tomography（OCT） Angiography after cataract surgery, to thoroughly evaluate the retinal state of diabetics after surgery, and to find out the relationship between postoperative complications occurred in retina and diabetes.

DETAILED DESCRIPTION:
In this study, we perform a completely comparison of retina state characteristic including the foveal avascular zone(FAZ),perifovea vessel density,parafovea vessel density,macular thickness,perifovea thickness,parafovea thickness in superficial and deep layers of retina with OCT Angiography after cataract surgery,and analysis on the differences of EGF,IFN-γ,IL-10,IL-12,IL-1β,IL-6,IL-8,IP-10,MCP-1,VEGF in aqueous humor before surgery between diabetic and non-diabetic patients and to explore the potential correlations between postoperative complications occurred in retina and diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age-related cataract and with willing to improve visual acuity by undergoing phacoemulsification and intraocular lens implantation surgery.
2. Type 2 diabetes diagnosis according to American Diabetes Association# Standards of Medical Care in Diabetes -2017(ADA, American Diabetes Association)
3. Willing to sign the consent form.

Exclusion Criteria:

1. having known maculopathy, proliferative diabetic retinopathy(PDR), diabetic macular edema.
2. with high myopia of spherical equivalent greater than -6.0 diopters or axial length (AXL) greater than 26 mm in either eye.
3. preexisting vein or artery occlusion,glaucoma, previous uveitis, a history of ocular trauma, laser treatment, intravitreal injections or intraocular surgeries.
4. patients who had complications during cataract surgery.

Elimination Criteria:

1. poor compliance
2. voluntary withdrawal
3. any other kind of situation that researchers consider not suitable for further study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population: Asian
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
OCT Angiography parameters | 3 months postoperatively
  comparison of vessel density in superficial and deep layers of retina between diabetic and non-diabetic patients with OCT Angiography.

SECONDARY OUTCOMES:
aqueous humor cytokines levels | intraoperatively.
  comparison the levels of cytokines from aqueous humor including EGF,IFN-γ，IL-10,IL-12,IL-1β，IL-6,IL-8,IP-10,MCP-1,VEGF between diabetic and non-diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China